CLINICAL TRIAL: NCT05825391
Title: Guided Versus Standard Antiplatelet Therapy in Intracranial Aneurysm Intervention With Stents: a Cluster Randomized Controlled Cohort Study
Brief Title: Guided Antiplatelet Therapy in Interventional Treatment of Intracranial Aneurysms
Acronym: GATITIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Chinese PLA General Hospital (Other); Beijing Chao Yang Hospital (Other); Peking University International Hospital (Other); Peking University First Hospital (Other); Hebei Medical University Third Hospital (Other); Tianjin Medical University General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Xinjian Yang
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Intracranial Aneurysm
Keywords: Intracranial Aneurysm; Interventional Therapy; Stent; Platelet; Ischemic Stroke; Bleeding Event
MeSH Terms: conditions — Intracranial Aneurysm; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: cluster randomized controlled cohort study
Who Masked: Outcomes Assessor
Masking Description: To ensure the reliability of the research results, a study committee consisting of 5 members will be formed. The committee comprised a 2-member data safety monitoring committee and a 3-member clinical event review committee. Each reported ischemic event and bleeding event were assessed independently by three members of the clinical event adjudication committee. These committee members were blinded to the treatment group assignments. Any disagreements were resolved by a third member of the clinical events adjudication committee. All five committee members reviewed and resolved any discrepancies through consensus.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Continue to use the center's original antiplatelet regimen: oral aspirin 100 mg and clopidogrel 75 mg daily
- test group (Experimental): Use a guided antiplatelet regimen based on LTA testing
  Interventions: Drug: Adjustment of Antiplatelet Drugs

INTERVENTIONS:
Drug: Adjustment of Antiplatelet Drugs — The maximum platelet aggregation rate induced by arachidonic acid (AA-MPA)≥20%, give aspirin 200mg qd. The maximum platelet aggregation rate induced by adenosine diphosphatase (ADP-MPA)≥36.4% for flow diversion, give ticagrelor 60mg bid. ADP-MPA≥42.9% for stent-assisted coil embolization，give ticagrelor 60mg bid. ADP-MPA<20%, give clopidogrel 37.5mg qd. The timing of drug adjustment should be at least 1 day before stent implantation, and the LTA testing should be performed again 48 hours after the drug adjustment. For patients whose ADP-MPA does not reach the normal range, a second antiplatelet drug adjustment should be performed: ticagrelor overdose: reduce to 45mg bid; ticagrelor resistance, increase to 90 mg bid.
  Arms: test group

SUMMARY:
The use of intracranial stents expands the possibilities for endovascular treatment of intracranial aneurysms and improves the success rate. However, it also increases the risk of ischemic complications in patients. The current standard dual antiplatelet regimen is considered crucial in reducing thrombotic events. Nevertheless, some patients exhibit resistance to antiplatelet drugs, which puts them at a higher risk of thrombotic events. In clinical practice, there is a lack of standardized platelet function testing and consensus on adjusting antiplatelet drug programs. This study conducted a multi-center, prospective cluster randomized controlled trial to investigate whether antiplatelet adjustment therapy guided by light transmittance aggregometry (LTA) detection can decrease the occurrence of ischemic events after stent implantation in patients with unruptured intracranial aneurysms. Additionally, the study aimed to establish a set of standardized antiplatelet regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unruptured intracranial aneurysms who received intracranial stenting,
2. Standard dualantiplatelet therapy for at least 5 days before stent implantation,
3. Patients aged 18-80,
4. on the day of registration patients with a Modified Rankin Scale lower than 2,
5. patients who agree and sign the consent form.

Exclusion Criteria:

1. Patients with recurrent aneurysms after interventional therapy or clipping therapy,
2. Patients with a history of allergy to aspirin, clopidogrel or ticagrelor,
3. Patients who used tirofiban prophylactically before surgery,
4. Possible active bleeding Patients with high blood pressure, such as symptomatic intracranial hemorrhage or active gastric ulcer; or patients with bleeding tendency or coagulation dysfunction,
5. Any abnormal platelet count (normal value is 100-300 × 10^9/L),
6. Patients using anticoagulants,
7. Pregnant or lactating women,
8. Suffering from liver disease, kidney disease, congestive heart failure, malignant tumors and other malignant diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-29 (Actual)

PRIMARY OUTCOMES:
Ischemic events | 30 days after stent implantation.
  ischemic stroke, transient ischemic stroke (TIA), stent thrombosis

OTHER OUTCOMES:
Bleeding events | 30 days after stent implantation.
  The primary safety endpoint was severe or life-threatening bleeding, moderate bleeding and minor bleeding, assessed according to the Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Arteries (GUSTO) classification.

CONTACTS AND LOCATIONS:
Overall Officials: Xinjian Yang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (2):
- China (2):
  - Beijing Tiantan hospital, Beijing, Beijing Municipality
  - Department of Neurosurgery, Beijing Tiantan Hospital., Beijing, Beijing Municipality

REFERENCES:
- [Result] Zhou Y, Li W, Wang C, Xie R, Zhu Y, Peng Q, Zhang L, Zhang H, Gu Y, Mu S, Liu J, Yang X. Roles of light transmission aggregometry and CYP2C19 genotype in predicting ischaemic complications during interventional therapy for intracranial aneurysms. Stroke Vasc Neurol. 2023 Aug;8(4):327-334. doi: 10.1136/svn-2022-001720. Epub 2023 Feb 6. PMID 36746550
- [Result] GUSTO investigators. An international randomized trial comparing four thrombolytic strategies for acute myocardial infarction. N Engl J Med. 1993 Sep 2;329(10):673-82. doi: 10.1056/NEJM199309023291001. PMID 8204123
- [Result] Easton JD, Saver JL, Albers GW, Alberts MJ, Chaturvedi S, Feldmann E, Hatsukami TS, Higashida RT, Johnston SC, Kidwell CS, Lutsep HL, Miller E, Sacco RL; American Heart Association; American Stroke Association Stroke Council; Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular Nursing; Interdisciplinary Council on Peripheral Vascular Disease. Definition and evaluation of transient ischemic attack: a scientific statement for healthcare professionals from the American Heart Association/American Stroke Association Stroke Council; Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular Nursing; and the Interdisciplinary Council on Peripheral Vascular Disease. The American Academy of Neurology affirms the value of this statement as an educational tool for neurologists. Stroke. 2009 Jun;40(6):2276-93. doi: 10.1161/STROKEAHA.108.192218. Epub 2009 May 7. PMID 19423857
- [Result] Sacco RL, Kasner SE, Broderick JP, Caplan LR, Connors JJ, Culebras A, Elkind MS, George MG, Hamdan AD, Higashida RT, Hoh BL, Janis LS, Kase CS, Kleindorfer DO, Lee JM, Moseley ME, Peterson ED, Turan TN, Valderrama AL, Vinters HV; American Heart Association Stroke Council, Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Council on Nutrition, Physical Activity and Metabolism. An updated definition of stroke for the 21st century: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Jul;44(7):2064-89. doi: 10.1161/STR.0b013e318296aeca. Epub 2013 May 7. PMID 23652265
- [Result] Gulliford MC, Adams G, Ukoumunne OC, Latinovic R, Chinn S, Campbell MJ. Intraclass correlation coefficient and outcome prevalence are associated in clustered binary data. J Clin Epidemiol. 2005 Mar;58(3):246-51. doi: 10.1016/j.jclinepi.2004.08.012. PMID 15718113
- [Derived] Zhou Y, Wang J, Li W, Liu J, Wang A, Zhang Y, Mu S, Xie R, Peng Q, Zhang L, Luo B, Zhao Y, Wang Y, Zhang Z, Lin Y, Zhang P, Zhang J, Li L, Yin X, Xiao F, Lin Y, Liu X, Bian Y, Wang S, Li J, Zhang X, Hasan DM, Krings T, Zhang H, Yang X. Guided Antiplatelet Therapy for Stent-Treated Intracranial Aneurysms: A Cluster-Randomized Trial. Radiology. 2025 Mar;314(3):e241509. doi: 10.1148/radiol.241509. PMID 40100020